CLINICAL TRIAL: NCT04312152
Title: Randomized, Placebo-controlled, Cross-over, Double-blind Study of a Metabolic Support Therapy With Q10 Ubiquinol and a Multivitamin B and E Complex in Two Cohorts of Patients With Idiopathic and Syndromic Autism (Phelan-McDermid Syndrome)
Brief Title: Q10 Ubiquinol in Autism Spectrum Disorder and in Phelan-McDermid Syndrome.
Acronym: Q10ASD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Antonio Persico (Other)
Collaborators: Associazione Italiana Sindrome di Phelan-McDermid (AISPHEM) (Unknown); University of Bari (Other)
Responsible Party: Sponsor-Investigator, Antonio Persico, Full Professor in Child & Adolescent Neuropsychiatry, University of Messina
Organization: University of Messina (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Q10_study_ASD
Record Dates: First submitted 2020-03-09; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Autism Spectrum Disorder; Phelan-McDermid Syndrome
Keywords: Ubiquinol-10; Coenzyme Q10; Autism; Mitochondria; Oxidative stress; Cognitive symptoms; Chromosome 22q13 3 deletion syndrome
MeSH Terms: conditions — Autism Spectrum Disorder; Telomeric 22q13 Monosomy Syndrome; Autistic Disorder; Neurobehavioral Manifestations | interventions — Vitamin E; Tocopherols

STUDY DESIGN:
Intervention Model Description: Each patient receives active compound [Q10 ubiquinol + Vit. E and polyvitamin B] for 4 months and placebo [Vit. E and B] for another 4 months. The total duration of the trial is 8 months. Half of the patients receive the active compound during months 1-4 and placebo during months 5-8, while the remaining half receives placebo during months 1-4 and active compound during months 5-8. Patients are assessed at T0, T4 and T8 mo. Administration of active compound and placebo is in double-blind.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, all care providers, investigators and outcome assessors are blind to treatment status, as well as patients and family. Three investigators with no contact with patients and families provide the appropriate blisters to patients. One investigator not involved in outcome assessment interacts with families for any question regarding the trial or medical issues, screening outcome assessors from contacts by families in between assessments (0-4-8 months). Families are requested to refrain from commenting their experience and trial outcome on social media.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PMS Placebo (Active Comparator): If body weight is up to 20 kg:
  * Vitamin E 30 mg b.i.d.
  * Multivitamin B complex b.i.d., including Vit. B1 (1.05 mg), Vit. B2 (1.2 mg), Niacin (9 mg), Pantothenic acid (4.5 mg), Vit. B6 (1.5 mg), Vit. B12 (4.5 mcg), Folic acid (0.1 mg), Biotin (0.1125 mg)
  If body weight is above 20 kg:
  * Vitamin E 30 mg b.i.d.
  * Multivitamin B complex b.i.d., including Vit. B1 (2.1 mg), Vit. B2 (2.4 mg), Niacin (18 mg), Pantothenic acid (9 mg), Vit. B6 (3 mg), Vit. B12 (9 mcg), Folic acid (0.2 mg), Biotin (0.225 mg)
  Interventions: Dietary Supplement: Vitamin E; Dietary Supplement: Multi-Vitamin B complex
- ASD Placebo (Active Comparator): If body weight is up to 20 kg:
  * Vitamin E 30 mg b.i.d.
  * Multivitamin B complex b.i.d., including Vit. B1 (1.05 mg), Vit. B2 (1.2 mg), Niacin (9 mg), Pantothenic acid (4.5 mg), Vit. B6 (1.5 mg), Vit. B12 (4.5 mcg), Folic acid (0.1 mg), Biotin (0.1125 mg)
  If body weight is above 20 kg:
  * Vitamin E 30 mg b.i.d.
  * Multivitamin B complex b.i.d., including Vit. B1 (2.1 mg), Vit. B2 (2.4 mg), Niacin (18 mg), Pantothenic acid (9 mg), Vit. B6 (3 mg), Vit. B12 (9 mcg), Folic acid (0.2 mg), Biotin (0.225 mg)
  Interventions: Dietary Supplement: Vitamin E; Dietary Supplement: Multi-Vitamin B complex
- PMS Active compound (Experimental): If body weight is up to 20 kg:
  * Q10 ubiquinol, 50 mg b.i.d.
  * Vitamin E 30 mg b.i.d.
  * Multivitamin B complex b.i.d., including Vit. B1 (1.05 mg), Vit. B2 (1.2 mg), Niacin (9 mg), Pantothenic acid (4.5 mg), Vit. B6 (1.5 mg), Vit. B12 (4.5 mcg), Folic acid (0.1 mg), Biotin (0.1125 mg)
  If body weight is above 20 kg:
  * Q10 ubiquinol, 100 mg b.i.d.
  * Vitamin E 30 mg b.i.d.
  * Multivitamin B complex b.i.d., including Vit. B1 (2.1 mg), Vit. B2 (2.4 mg), Niacin (18 mg), Pantothenic acid (9 mg), Vit. B6 (3 mg), Vit. B12 (9 mcg), Folic acid (0.2 mg), Biotin (0.225 mg)
  Interventions: Dietary Supplement: Q10 Ubiquinol; Dietary Supplement: Vitamin E; Dietary Supplement: Multi-Vitamin B complex
- ASD Active compound (Experimental): If body weight is up to 20 kg:
  * Q10 ubiquinol, 50 mg b.i.d.
  * Vitamin E 30 mg b.i.d.
  * Multivitamin B complex b.i.d., including Vit. B1 (1.05 mg), Vit. B2 (1.2 mg), Niacin (9 mg), Pantothenic acid (4.5 mg), Vit. B6 (1.5 mg), Vit. B12 (4.5 mcg), Folic acid (0.1 mg), Biotin (0.1125 mg)
  If body weight is above 20 kg:
  * Q10 ubiquinol, 100 mg b.i.d.
  * Vitamin E 30 mg b.i.d.
  * Multivitamin B complex b.i.d., including Vit. B1 (2.1 mg), Vit. B2 (2.4 mg), Niacin (18 mg), Pantothenic acid (9 mg), Vit. B6 (3 mg), Vit. B12 (9 mcg), Folic acid (0.2 mg), Biotin (0.225 mg)
  Interventions: Dietary Supplement: Q10 Ubiquinol; Dietary Supplement: Vitamin E; Dietary Supplement: Multi-Vitamin B complex

INTERVENTIONS:
Dietary Supplement: Q10 Ubiquinol — Q10 Ubiquinol (50 or 100 mg b.i.d. depending on body weight) in capsules containing also Vit. E and Vit. B complex, as described above. Capsules can be opened and the content drunk or chewed, if children have difficulties with swallowing capsules.
  Arms: ASD Active compound; PMS Active compound
Dietary Supplement: Vitamin E — Vitamin E (30 mg b.i.d. regardless of body weight) in capsules containing also Vit. B complex, and, in the active arms, Q10 ubiquinol. Capsules can be opened and the content drunk or chewed, if children have difficulties with swallowing capsules.
  Other Names: tocopherols
Dietary Supplement: Multi-Vitamin B complex — Multi-Vitamin B complex including Vit. B1, B2, B3, B5, B6, B8, B9, and B12, in capsules containing also Vit. E and, in the active arms, Q10 ubiquinol. Capsules can be opened and the content drunk or chewed, if children have difficulties with swallowing capsules.

SUMMARY:
This double-blind, cross-over, randomized, controlled trial (RCT) has the aim of evaluating the effectiveness of a metabolic support therapy in two cohorts of patients with idiopathic Autism Spectrum Disorder or Phelan-McDermid syndrome, commonly associated with syndromic autism. Each patient will receive Q10 ubiquinol + Vit. E and B for 4 months and only Vit. E and B for 4 months in a double-blind, cross-over design. Primary outcome measures of efficacy include Vineland Adaptive Behavior Scales, Childhood Autism Rating Scale, Clinical Global Impression-Improvement and Visual Analog Scales; secondary outcome measures include several questionnaires and tests of autism, cognitive function, problem behaviors, quality of life, communication and comorbid disorders, as well as measures of oxidative stress.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a clinically and genetically heterogeneous collection of different conditions, sharing socio-communicative deficits, repetitive behaviors, restricted interests, and dysfunctional sensory processing. Currently there are no pharmaceutical compounds effective on core ASD symptoms. Enhanced oxidative stress and mitochondrial dysfunction represent one of the most replicated abnormalities detected both systemically and in the Central Nervous System (CNS) of autistic individuals. Abnormalities in redox parameters are significantly correlated with the severity of autistic behaviors. Although oxidative stress usually represents the consequence and not the primary cause of ASD, reduced ATP production and oxidative damage can seemingly contribute an additional burden to the dysfunction directly produced by ASD-causing genetic or epigenetic defects. Importantly, redox abnormalities have been detected also in young autistic children and are not correlated with age. Therefore, enhanced oxidative stress and mitochondrial dysfunction represent an ASD-related "state-dependent" characteristic present in a consistent number of autistic individuals regardless of their age and of their specific underlying pathogenetic underpinnings. Sustaining mitochondrial function while controlling redox imbalance thus represents a viable "indirect" therapeutic approach, potentially able to ameliorate behavioral and neuropsychological deficits in many autistic individuals.

Coenzyme Q10 (CoQ10, ubiquinone or ubiquinol) is a lipid soluble compound present in the majority of living cells. By increasing energy production and antioxidant capacity, CoQ10 is predicted to limit the damage generated by the neuroinflammation and excitotoxicity well documented in ASD brains, ultimately leading to excessive neuritic pruning and/or cell apoptosis. Administration of Q10 ubiquinol to autistic children, as frequently prescribed to children with mitochondrial disorders, yielded promising results with an extremely low incidence and minor impact of side effects in two open trials and in three RCTs involving numerous other active compounds. In the present RCT, each patient will receive Q10 ubiquinol (50-100 mg b.i.d.) + Vit. E (60 mg/die) and polyvitamin B for 4 months and only Vit. E and B for another 4 months (total duration 8 months) in a double-blind, cross-over design. The focused co-administration of Q10 ubiquinol with only two known antioxidants, vitamin E and a multivitamin B complex, is designed to synergistically boost the increase in energy production and cell protection viewed as deriving primarily from Q10 ubiquinol administration. This study was also designed to overcome two limitations present in previous RCTs evaluating the effects of Q10 Ubiquinone (precursor of Q10 ubiquinol) in ASD children and adults: (a) The administration of a very limited number of active compounds, as compared to cocktails containing many active substances, allows to focus here on the efficacy of Q10 ubiquinol; (b) the administration of Q10 ubiquinol, rather than its precursor Q10 ubiquinone, avoids the potential risk of reduced response due to pharmacokinetic interference with the biotransformation of the precursor into the active compound.

This trial addresses the efficacy of Q10 ubiquinol, paired with Vit. E and B, not only in "idiopathic" ASD, but also in "syndromic" ASD, using Phelan-McDermid syndrome (PMS) as a paradigm. PMS, also known as chromosome 22q13.3 deletion syndrome, represents one of the most studied syndromic forms of ASD. It is characterized by autism in as many as 70-80% of deletion carriers, in addition to early onset severe muscle hypotonia, developmental delay, facial dysmorphisms, absence of spoken language or severe language development disorder. Deletions or mutations of the SHANK3 gene, encoding a synaptic scaffold protein critical to glutamatergic synapse function, are primarily responsible for the syndrome, although larger 22q13.3 deletions encompass additional disease genes.

This study shall include up to 140 patients with idiopathic ASD and 60 patients with PMS. The study design of this RCT was balanced, so that half of the patients with ASD or PMS will receive Q10 ubiquinol during the first 4 months, and the remaining half will receive Q10 ubiquinol during the second 4 months. The purpose of this balancing is to observe not only whether Q10 ubiquinol produces and improvement in primary and secondary measures, but also if this improvement is sustained over time despite Q10 discontinuation or requires continued Q10 administration. In addition to clinical and psychometric parameters, oxidative stress will be measured at baseline and after 4 and 8 months, by drawing 8-10 ml of blood, isolating leukocytes by Ficoll gradient and assessing (a) protein carbonylation levels by oxyblot; (b) the activity of mitochondrial respiratory chain complexes normalized by citrate synthase activity; (c) the expression levels of mitochondrial respiratory chain complexes measured by Western-Blotting.

ELIGIBILITY:
Inclusion Criteria:

1. Both parents or a legally authorized patient representative (LAR) must provide written informed consent. The parents and guardian must be able to understand and comply with the experimental protocol;
2. Subjects of both sexes, aged between 2 and 40 years old, may be included in the study;
3. The subject must meet DSM-5 criteria for a primary diagnosis of Autism Spectrum Disorder (idiopathic autism) or carry a documented deletion of human chromosome 22q13.33 or mutation in the SHANK3 gene (Phelan-McDermid Syndrome);
4. Subjects with idiopathic autism must pass the threshold score for Autism of the Autism Diagnostic Observation Schedule;
5. Baseline Children's Global Assessment Scale score must be between 45 and 59;
6. Patients treated with psychoactive drugs (neuroleptics, antiepileptics, etc.) are enrolled only if the treatment and dosage of these drugs has been constant for at least 3 months prior to enrollment in the trial and is kept constant throughout the 8-month duration of the trial;
7. Patients undergoing any kind of behavioral intervention must have must have started the intervention at least 3 months prior to enrollment and the intervention must remain unchanged throughout the 8-month duration of the trial;
8. The patient is able to swallow the capsule or his/her parents are available to open it and administer immediately its content in a small quantity of juice or soft-drink.

Exclusion Criteria:

Patients who meet any of the following criteria will not be recruited in the study:

1. Patients with autism secondary to known genetic syndromes other than Phelan-McDermid syndrome (for example, Rett syndrome, fragile-X syndrome, etc.);
2. Presence of brain malformations or major structural anomalies visible by magnetic resonance imaging;
3. Patients with autism secondary to epileptic encephalopathy or with idiopathic autism comorbid with seizures more frequent than one episode every 6 months despite ongoing antiepileptic drug therapy;
4. Patients with autism accompanied by marked facial dysmorphism and/or congenital malformations;
5. Patients treated with anticoagulants;
6. Patients with serious medical illnesses (chronic renal disease, severe liver disease, cardiovascular disorders, uncontrolled hypertension with systolic pressure values> 170 and diastolic pressure> 100 mm Hg, malignant tumors, HIV infection);
7. Patients with a history of acute cerebrovascular episodes;
8. Patients with a history of stomach bleeding or active peptic ulcer;
9. Patients with documented allergy, hypersensitivity or intolerance to one of the excipients of the experimental or comparative product.

Trial interruption criteria:

1. Patients whose medical conditions require starting treatment with anticoagulants.
2. Patients with severe medical conditions starting during the 8-month duration of the trial.
3. Patients who undergo a change in psychopharmacological or behavioral treatment during the 8-month duration of the trial.

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-03-09 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Vineland Adaptive Behavior Scales scores | At 0, 4 and 8 months (pre- and post-treatment after each arm)
  The Vineland Adaptive Behavior Scales are a standardized semi-structured interview to measure adaptive behavior, among the most sensitive to change in autism research. Standard scores have a mean of 100 and a standard deviation of 15.
Change in Childhood Autism Rating Scale score | At 0, 4 and 8 months (pre- and post-treatment after each arm)
  The Childhood Autism Rating Scale is a clinical rating scale for the trained clinician to rate the presence and severity of signs and symptoms of ASD by direct observation of the child. Scores can range from 15 to 60: below 30, non-autistic; 30-36.5, mild to moderate autism; 37-60, severe autism.
Change in Clinical Global Impression of Improvement scale scores between experimental and active comparator arms. | 4 and 8 months (record once at the end of each arm)
  The Clinical Global Impression of Improvement scale is a 7 point scale for the clinician to quantify illness severity, patient improvement/worsening and treatment side effects. Scores recorded at the end of the experimental and active comparator arms will be contrasted within-subject.
Change in Visual Analog Scales scores | At 0, 4 and 8 months (pre- and post-treatment after each arm)
  16 visual analog scales have been created to measure all DSM-5 items included in the ASD diagnosis, as well as other cognitive and motor functions often affected in ASD. Scores measure the increasing severity of signs and symptoms on a 0-10 scale.

SECONDARY OUTCOMES:
Children's Global Assessment Scale | At 0, 4 and 8 months (pre- and post-treatment after each arm)
  The Children's Global Assessment Scale provides a global measure of level of functioning in children and adolescents. The measure provides a single rating on a 0-100 scale, with higher scores indicating better functioning.
Social Responsiveness Scale | At 0, 4 and 8 months (pre- and post-treatment after each arm)
  65-item questionnaire used to assess social impairment, communication deficits and repetitive behaviors in children and adolescents 4-18 years old. Autism is severe, moderate, or mild when T-scores are above 75, 66-75, or 60-65, respectively. Scores below 60 are not clinically significant.
Repetitive Behaviors Scale - Revised | At 0, 4 and 8 months (pre- and post-treatment after each arm)
  44-item questionnaire used to assess repetitive behaviors. Filled by parents for children 6-17 years old. Behaviors are rated on a 0-3 scale to measure increasing symptom severity, as does the overall global score ranging 0-100.
Aberrant Behavior Checklist | At 0, 4 and 8 months (pre- and post-treatment after each arm)
  58-item questionnaire used to assess problem behaviors with parents or guardians. Behaviors are rated on a 0-3 scale to measure increasing symptom severity.
Short Sensory Profile | At 0, 4 and 8 months (pre- and post-treatment after each arm)
  38-item questionnaire filled by caregivers to assess the sensory profile of patients, including sensory processing, modulation, and behavioral/emotional responses. The overall score ranges from 0 to 190, with lower scores reflecting greater symptom severity.
Conners' Parent Rating Scale-Revised | At 0, 4 and 8 months (pre- and post-treatment after each arm)
  48-item rating scale used to evaluate through parental reports the presence and intensity of childhood hyperactivity/inattention, impulsivity and externalizing behaviors. Each item is rated on a 0-3 scale to reflect increasing symptom severity.
Child Behavior Checklist | At 0, 4 and 8 months (pre- and post-treatment after each arm)
  The Child Behavior Checklist/6-18 provides ratings for 20 competence and 120 behavioral problem items of youth aged 6-18 years old by parental report. Each item is scored 0-2, to reflect symptom severity or frequency. Standard scores are scaled so that 50 is average for the youth's age and gender, with a standard deviation of 10 points.
Intellectual Quotient | At 0, 4 and 8 months (pre- and post-treatment after each arm)
  Intellectual quotient measured as a standardized score with population mean 100 and standard deviation 15, using one cognitive test per subject, chosen depending on age and language development (either Griffiths Developmental Rating Scales, Wechsler Intelligence Scale for Children - Fourth Edition, or Leiter III).
The Quality of Life in Autism Questionnaire | At 0, 4 and 8 months (pre- and post-treatment after each arm)
  A questionnaire used to assess parental quality of life either broadly (part A, 28 items, score range 28-140) or specifically related to the autism present in their offspring (part B, 20 items, score range 20-100). Total score range 48-240, with higher scores indicating better quality of life.
The World Health Organization's Quality of Life Questionnaire | At 0, 4 and 8 months (pre- and post-treatment after each arm)
  A questionnaire used to assess parental quality of life in four domains: physical, psychological, social, and environmental. The score can range from 15 to 105, with a higher score being indicative of a higher quality of life.
Measurement of protein carbonylation level as a marker of oxidative stress in leukocytes. | Blood drawn at 0, 4 and 8 months (pre-and post-treatment after each arm).
  Blood drawing, isolation of leukocytes by Ficoll gradient and measurement of protein carbonylation by oxyblot.
Measurement of the activity of mitochondrial respiratory chain complexes. | Blood drawn at 0, 4 and 8 months (pre-and post-treatment after each arm).
  Blood drawing, isolation of leukocytes by Ficoll gradient and measurement of the activity of mitochondrial respiratory chain complexes normalized by citrate synthase activity.
Measurement of expression levels of mitochondrial respiratory chain complexes. | Blood drawn at 0, 4 and 8 months (pre-and post-treatment after each arm).
  Blood drawing, isolation of leukocytes by Ficoll gradient and measurement of the expression levels of mitochondrial respiratory chain complexes by Western-Blotting.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio M. Persico, MD, Principal Investigator — University of Messina
Locations (1):
- Interdipartimental Program "Autismo 0-90" at "G. Martino" Universitary Hospital, Messina, ME, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders. In: Association AP, editor. Fifth Edition ed: American Psychiatric Publishing, Arlington; 2013.
- [Background] Persico AM, Arango C, Buitelaar JK, Correll CU, Glennon JC, Hoekstra PJ, Moreno C, Vitiello B, Vorstman J, Zuddas A; European Child and Adolescent Clinical Psychopharmacology Network. Unmet needs in paediatric psychopharmacology: Present scenario and future perspectives. Eur Neuropsychopharmacol. 2015 Oct;25(10):1513-31. doi: 10.1016/j.euroneuro.2015.06.009. Epub 2015 Jun 20. PMID 26166453
- [Background] Kalayci M, Unal MM, Gul S, Acikgoz S, Kandemir N, Hanci V, Edebali N, Acikgoz B. Effect of coenzyme Q10 on ischemia and neuronal damage in an experimental traumatic brain-injury model in rats. BMC Neurosci. 2011 Jul 29;12:75. doi: 10.1186/1471-2202-12-75. PMID 21801363
- [Background] Kumari S, Mehta SL, Milledge GZ, Huang X, Li H, Li PA. Ubisol-Q10 Prevents Glutamate-Induced Cell Death by Blocking Mitochondrial Fragmentation and Permeability Transition Pore Opening. Int J Biol Sci. 2016 Apr 27;12(6):688-700. doi: 10.7150/ijbs.13589. eCollection 2016. PMID 27194946
- [Background] Duberley KE, Heales SJ, Abramov AY, Chalasani A, Land JM, Rahman S, Hargreaves IP. Effect of Coenzyme Q10 supplementation on mitochondrial electron transport chain activity and mitochondrial oxidative stress in Coenzyme Q10 deficient human neuronal cells. Int J Biochem Cell Biol. 2014 May;50:60-3. doi: 10.1016/j.biocel.2014.02.003. Epub 2014 Feb 15. PMID 24534273
- [Background] Rossignol DA, Frye RE. Evidence linking oxidative stress, mitochondrial dysfunction, and inflammation in the brain of individuals with autism. Front Physiol. 2014 Apr 22;5:150. doi: 10.3389/fphys.2014.00150. eCollection 2014. PMID 24795645
- [Background] Frustaci A, Neri M, Cesario A, Adams JB, Domenici E, Dalla Bernardina B, Bonassi S. Oxidative stress-related biomarkers in autism: systematic review and meta-analyses. Free Radic Biol Med. 2012 May 15;52(10):2128-41. doi: 10.1016/j.freeradbiomed.2012.03.011. Epub 2012 Apr 18. PMID 22542447
- [Background] Adams JB, Baral M, Geis E, Mitchell J, Ingram J, Hensley A, Zappia I, Newmark S, Gehn E, Rubin RA, Mitchell K, Bradstreet J, El-Dahr JM. The severity of autism is associated with toxic metal body burden and red blood cell glutathione levels. J Toxicol. 2009;2009:532640. doi: 10.1155/2009/532640. Epub 2009 Aug 26. PMID 20107587
- [Background] Ghezzo A, Visconti P, Abruzzo PM, Bolotta A, Ferreri C, Gobbi G, Malisardi G, Manfredini S, Marini M, Nanetti L, Pipitone E, Raffaelli F, Resca F, Vignini A, Mazzanti L. Oxidative Stress and Erythrocyte Membrane Alterations in Children with Autism: Correlation with Clinical Features. PLoS One. 2013 Jun 19;8(6):e66418. doi: 10.1371/journal.pone.0066418. Print 2013. PMID 23840462
- [Background] Adams JB, Holloway C. Pilot study of a moderate dose multivitamin/mineral supplement for children with autistic spectrum disorder. J Altern Complement Med. 2004 Dec;10(6):1033-9. doi: 10.1089/acm.2004.10.1033. PMID 15673999
- [Background] Adams JB, Audhya T, McDonough-Means S, Rubin RA, Quig D, Geis E, Gehn E, Loresto M, Mitchell J, Atwood S, Barnhouse S, Lee W. Effect of a vitamin/mineral supplement on children and adults with autism. BMC Pediatr. 2011 Dec 12;11:111. doi: 10.1186/1471-2431-11-111. PMID 22151477
- [Background] Adams JB, George F, Audhya T. Abnormally high plasma levels of vitamin B6 in children with autism not taking supplements compared to controls not taking supplements. J Altern Complement Med. 2006 Jan-Feb;12(1):59-63. doi: 10.1089/acm.2006.12.59. PMID 16494569
- [Background] Palmieri L, Persico AM. Mitochondrial dysfunction in autism spectrum disorders: cause or effect? Biochim Biophys Acta. 2010 Jun-Jul;1797(6-7):1130-7. doi: 10.1016/j.bbabio.2010.04.018. Epub 2010 May 9. PMID 20441769
- [Background] Gvozdjakova A, Kucharska J, Ostatnikova D, Babinska K, Nakladal D, Crane FL. Ubiquinol improves symptoms in children with autism. Oxid Med Cell Longev. 2014;2014:798957. doi: 10.1155/2014/798957. Epub 2014 Feb 23. PMID 24707344
- [Background] Mousavinejad E, Ghaffari MA, Riahi F, Hajmohammadi M, Tiznobeyk Z, Mousavinejad M. Coenzyme Q10 supplementation reduces oxidative stress and decreases antioxidant enzyme activity in children with autism spectrum disorders. Psychiatry Res. 2018 Jul;265:62-69. doi: 10.1016/j.psychres.2018.03.061. Epub 2018 Apr 4. PMID 29684771
- [Background] Adams JB, Audhya T, Geis E, Gehn E, Fimbres V, Pollard EL, Mitchell J, Ingram J, Hellmers R, Laake D, Matthews JS, Li K, Naviaux JC, Naviaux RK, Adams RL, Coleman DM, Quig DW. Comprehensive Nutritional and Dietary Intervention for Autism Spectrum Disorder-A Randomized, Controlled 12-Month Trial. Nutrients. 2018 Mar 17;10(3):369. doi: 10.3390/nu10030369. PMID 29562612
- [Background] Harony-Nicolas H, De Rubeis S, Kolevzon A, Buxbaum JD. Phelan McDermid Syndrome: From Genetic Discoveries to Animal Models and Treatment. J Child Neurol. 2015 Dec;30(14):1861-70. doi: 10.1177/0883073815600872. Epub 2015 Sep 8. PMID 26350728